CLINICAL TRIAL: NCT02492321
Title: A Multi-Center, Randomized, Double-Masked, Vehicle-Controlled Evaluation of the Efficacy, Safety, and Tolerability of EBI-005 in Subjects With Moderate to Severe Ocular Allergic Conjunctivitis
Brief Title: A Multi-Center Environmental Study for the Treatment of Moderate to Severe Ocular Allergic Conjunctivitis
Acronym: EBI-005-AC-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eleven Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EBI-005-AC-2
Record Dates: First submitted 2015-07-02; First posted 2015-07-08 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Allergic Conjunctivitis (AC)
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — EBI-005

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EBI-005 (Active Comparator): Drug: EBI-005 The investigational drug EBI-005, is an intervention to one of two study arms: 5 mg/mL topical administered 3 times per day
  Interventions: Drug: EBI-005
- Vehicle (Placebo Comparator): Placebo Comparator: One of two study arms: placebo topical administered 3 times per day
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: EBI-005
  Arms: EBI-005
Drug: Placebo Comparator
  Arms: Vehicle

SUMMARY:
This is a Phase III multi-center, double-masked, vehicle-controlled, randomized, parallel group study evaluating the efficacy, safety and tolerability of EBI-005 as compared to vehicle given as a topical ophthalmic solution in each eye to subjects with moderate to severe allergic conjunctivitis (AC) three times daily for 4 weeks.

Approximately 250 subjects at approximately 8 centers in the US will be screened and enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent and any authorization required by local law (e.g., Protected Health Information waiver) prior to performing any study procedures;
* Are ≥18 years of age;
* Have a positive history of ocular allergies during ragweed pollen season;
* Have signs and symptoms of allergic conjunctivitis in both eyes;
* If female and of child-bearing potential, she must not be pregnant or lactating

Exclusion Criteria:

* Have signs of ocular infection;
* Have a known history of alcohol or drug abuse;
* Have been exposed to an investigational drug or device within 30 days of the study;
* Have planned surgery (ocular or systemic) during the trial period or within 30 days after

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Morning ocular itching diary scores | 14 days
  To evaluate the efficacy of EBI-005 as compared to vehicle-control in the treatment of ocular itching associated with allergic conjunctivitis during ragweed pollen season.

SECONDARY OUTCOMES:
Late afternoon ocular itching diary scores | 14 days
  The key secondary endpoints are to evaluate the efficacy of EBI-005 as compared to vehicle-control in the treatment of ocular itching associated with allergic conjunctivitis during ragweed pollen season
Evening ocular itching diary scores | 14 days
  The key secondary endpoints are to evaluate the efficacy of EBI-005 as compared to vehicle-control in the treatment of ocular itching associated with allergic conjunctivitis during ragweed pollen season

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldstein, MD, Study Director — Eleven Biotherapeutics
Locations (11):
- United States (11):
  - Morrow, Georgia
  - Louisville, Kentucky
  - Andover, Massachusetts
  - Investigational Site, Quincy, Massachusetts
  - Investigational Site, St Louis, Missouri
  - Charlotte, North Carolina
  - Investigational Site, Cincinnati, Ohio
  - Investigational Site, Mason, Ohio
  - Investigational Site, Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - San Antonio, Texas